CLINICAL TRIAL: NCT06374823
Title: The Impact of Multiple Electrolytes Injection (II) and Normal Saline on Hyperchloremia in Severe Hemorrhagic Stroke Patients: A Prospective, Multicenter, Open-label, Randomized Controlled Study
Brief Title: Multiple Electrolytes Injection (II) and Normal Saline on Hyperchloremia in Severe Hemorrhagic Stroke
Acronym: MERIT
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jian-Xin Zhou, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023-020-002
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Critical Care; Hyperchloremia; Hemorrhagic Stroke
Keywords: Saline; Crystalloid Solution
MeSH Terms: conditions — Hemorrhagic Stroke | interventions — Saline Solution; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multiple Electrolyte (Experimental): Multiple Electrolytes Injection(II): contains sodium chloride 6.799g, potassium chloride 0.2984g, calcium chloride 0.3675g, magnesium chloride 0.2033g, sodium acetate 3.266g, L-malic acid 0.671, sodium hydroxide 0.200g per 1000mL.
  Interventions: Drug: Multiple Electrolyte
- Normal Saline (Active Comparator): Sodium chloride injection: contains sodium chloride 9.0g per 1000mL.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Multiple Electrolyte — Patients who are randomized to multiple electrolyte group will be receiving Multiple Electrolytes injection II for 72 hours continously after inrollment as maintence and rescutation fluids. Infusion speed and volume will be determained by physicians.
  Other Names: Multiple Electrolytes injection II
  Arms: Multiple Electrolyte
Drug: Normal Saline — Patients who are randomized to normal saline group will be receiving Sodium Chloride injection for 72 hours continously after inrollment as maintence and rescutation fluids. Infusion speed and volume will be determained by physicians.
  Other Names: Sodium Chloride injection
  Arms: Normal Saline

SUMMARY:
Normal saline (0.9% sodium chloride), a classical crystalloid solution, is widely used to maintain fluid balance, volume resuscitation and dilute drugs during clinical practice. However, the chloride concentration of normal saline (154mmol/L) is much higher than human plasma, and a large amount of infusion may lead to iatrogenic hyperchloremia in ICU patients. In contrast, the concentrations of Multiple electrolytes II is more similar to those of plasma and is considered to be a better fluid choice than normal saline.

DETAILED DESCRIPTION:
Fluid therapy remains an important part of the treatment and management of critically ill patients. An everyday fluid intake can be simplely divided into: resuscitation fluid, maintenance fluid, nutrition, blood products, drugs and drug carriers. Daily resuscitation and maintenance fluids can account for 31.2% of the total fluid intake and increase during the first 3 days of admission, up to 58.1%, resulting in heavy sodium and chloride loads.

Among them, normal saline (0.9% sodium chloride), a classical crystalloid solution, is widely used to maintain fluid balance, volume resuscitation and dilute drugs. However, the chloride concentration of normal saline (154mmol/L) is much higher than that of human plasma, and a large amount of infusion may lead to iatrogenic hyperchloremia in ICU patients. Hyperchloremia is thought to cause acidosis, decrease in the glomerular filtration rate, impaired renal function, and even mortality. In contrast, the concentrations of balanced crystalloid solutions are more similar to those of plasma and is considered to be a better fluid choice than normal saline.

Hemorrhagic Stroke, which includes spontaneous cerebral hemorrhage and subarachnoid hemorrhage (SAH), is characterized by high mortality and disability. According to the latest studies, there are approximately 1.7 million new hemorrhagic strokes in China each year, and hemorrhagic strokes account for only 30% of all new stroke cases, but 60% of stroke deaths. There is a lack of relevant research on fluid recommendation for this population. One study of subarachnoid hemorrhage suggested that saline caused hyperchloremia, hypertonia, and positive fluid balance over 1500 mL in a large number of patients early after SAH.

Multiple electrolytes II, as a new isotonic balanced salt solution, contains a variety of cations (sodium, potassium, calcium, magnesium) and a lower chloride concentration than normal saline. A study of 30 patients demonstrated that it improved acid-base balance when used in neurosurgery. It may be a new alternative to sodium chloride solution.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of hemorrhagic stroke (cerebral hemorrhage, intraventricular hemorrhage, or subarachnoid hemorrhage confirmed by CT or MRI, except for subdural or extradural hemorrhage caused by tramma)
* Patients requiring fluid therapy
* Patients over 18 years old

Exclusion Criteria:

* Hemorrhage onset more than 72hours
* Preexisting hyperchloremia(blood chloride > 110mmol/L)
* Presence of hypothalamic disease or cerebral salt wasting syndrome
* Patients who can eat by themselves
* Patients receiving routine RRT
* Patients with known allergic or adverse reactions to the liquid used
* Patients with organ failure (such as heart failure, renal failure, liver failure) or end-stage disease
* Patients with autoimmune diseases, inflammatory diseases, metabolic diseases and blood diseases
* Patients with serious heart disease or arrhythmia
* Patients who are expected to have difficulty complying with the study plan or collecting data completely
* Pregnant or lactating women
* No informed consent was signed
* Patients participating in other clinical trials
* Other conditions deemed by the investigator to be ineligible for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Hyperchloremia | At 24 hours, 48 hours, 72 hours after enrollment
  The incidence of hyperchloremia

SECONDARY OUTCOMES:
Hyperchloremia acidosis | At 24 hours, 48 hours, 72 hours after enrollment
  Incidence of hyperchloremia acidosis
Plasma osmolality | At 24 hours, 48 hours, 72 hours after enrollment
  Plasma osmolality calculate by algorithm
AKI | recorded till day 7 after enrollment
  Incidence of acute kidney injury
RRT | recorded till day 7 after enrollment
  Incidence of new renal replacement therapy
hospital length of stay | recorded at discharge or 28 days after enrollment
  hospital length of stay
ICU length of stay | recorded at ICU discharge or 28 days after enrollment
  ICU length of stay
hospitalization expense | recorded at discharge or 28 days after enrollment
  hospitalization expense

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Xin Zhou, MD, Principal Investigator — Capital Medical University
Locations (1):
- Beijing Shijitan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No